CLINICAL TRIAL: NCT01294046
Title: Electrical Stimulation of the Sphenopalatine Ganglion for the Treatment of Migraine Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Autonomic Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE Number : G100007
Record Dates: First submitted 2011-02-04; First posted 2011-02-11 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Migraine Headache
Keywords: Episodic migraine headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep brain stimulation of SPG for migraine (Experimental): Electrical SPG for Treatment of Migraine
  Interventions: Device: Deep Brain Stimulation of SPG for Migraine

INTERVENTIONS:
Device: Deep Brain Stimulation of SPG for Migraine — Deep Brain Stimulation of SPG for Migraine
  Other Names: Medtronic 37702 PrimeAdvanced™

SUMMARY:
This investigation will gather information about a procedure called sphenopalatine ganglion (SPG) stimulation, and its appropriateness, safety, and efficacy as a treatment for those who suffer migraine headaches which may result in chronic severe disability. The SPG is a small collection of nerve cells in the head, and is located near the base of the nose on either side. Participation involves the surgical implantation of an electrode (small electrical conductor) over the sphenopalatine ganglion. The electrode is connected to a stimulator which will enable treatment for migraine headaches. Tiny electrical current is delivered to the stimulator device by an internal pulse generator implanted in the area at the top of the chest, to stop the migraine headaches. The implant system will be controlled with a wireless remote provided after the implant procedure.

Participation will record headache diaries throughout the study, which will last approximately 8½ months, and a yearly visit annually for five years.

DETAILED DESCRIPTION:
This application proposes a clinical study of electrical stimulation of the sphenopalatine ganglia (SPG) as a treatment for up to three individuals with episodic migraine headache. The present study is aimed at obtaining pilot data to guide a future controlled trial of this treatment modality. The study population will include individuals suffering from episodic migraine headaches with chronic severe disability, as demonstrated by the Migraine Disability Assessment Questionnaire (Lipton, 2000) and Headache Impact Test short form (HIT-6™) (Kosinski, 2003).

The treatment involves implantation of an electrode into the SPG. The electrode is connected subcutaneously to an infraclavicular stimulator (PrimeAdvanced™ 37702 Multi-program Neurostimulator System, Medtronic Inc., Minneapolis MN). Proper electrode placement will be verified using anatomic and physiologic techniques. Participants will receive the Medtronic Model 3389 or 3387 lead, or Medtronic subcompact lead Model 3776-45, 3776-60, or 3776-75. Stimulation will be delivered in a range of frequencies from 20 to 130 Hz, and pulse width from 60 to 450 μsec, and a titrated voltage. The voltages used for chronic stimulation may range up to the pulse generator maximum of 10.5 volts but are anticipated to generally be below 3 volts, keeping below the 30 µcoulomb/cm² charge density safety limit, and below the threshold for adverse stimulation-related effects. The minimum number of contacts on the quadripolar leads will be activated as necessary to produce a response.

The Prime Advanced neurostimulator to be used in this study allows the clinician to set all stimulation parameters including the maximum allowable amplitude. It is our responsibility to assure that appropriate stimulation parameters are used to result in appropriate electrical exposure charge density) below a 30 µC/cm2/phase limit. As is done with commercially available neurostimulators, during this study, we will utilize the charts presented in Figures 1 and 2 below to assist in selection of programming parameters, and this programming will be maintained by software controls within the neurostimulator.

For this exploratory study of 3 patients, the maximum electrical stimulating parameters, resulting electrical exposure (e.g., charge density), will be determined using the methods described above. It is our responsibility to assure that safe stimulation parameters are used at all times and that the maximum settings do not exceed the safety limits. Our plan is to begin with lead 3776 if possible, because it does not require an extra extension, but we would use 3387 or 3389 if clinically indicated.

The proposed study is a physician-sponsored research investigation of three patients, and the attention to stimulation parameters will be much greater than can be expected for a commercially released product. It is our responsibility within this investigational study to insure the selected stimulation parameters do not exceed the safety limit of 30μC/cm2/phase. Patients participating in the study will only be able to lower stimulation amplitudes, thereby keeping stimulation parameters BELOW any clinician set maximum. The only programs available to or accessible by the patients will maintain the previously described parameter set limitations. Thus, the programming of the Implantable Programmable Generator (IPG) will keep the three patients from stimulating outside or above the set and safe parameters.

The primary outcome measures for assessing the efficacy of migraine treatment will be a subject reported daily diary noting frequency and intensity of headaches. During this investigation we will obtain preliminary controlled data on the safety and efficacy of SPG stimulation for migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Subject has onset of migraine headache occurring before age 60.
3. Subject has been diagnosed with migraine headache with or without aura, according to the 2004 IHS criteria 1.1 and 1.2.
4. Subject reports a HIT-6 score of >56, a MIDAS score of >20 and/or a failure of adequate and appropriate previous migraine treatment.
5. Subject has carried the diagnosis of migraine for at least 6 months prior to enrollment.
6. Subject has had at least three migraine headache attacks per month.
7. Subject has had at least three headache days (migraine or non-migraine) per month and maintains this requirement during the baseline period on diary.
8. Subject is able to distinguish migraine headache attacks as discrete from other headaches (i.e., tension-type headaches).
9. Subject has the ability to read, comprehend and legibly and reliably record information as required by the protocol.
10. Subject is able to provide written informed consent prior to participation in the study.
11. Subject agrees to not participate in supplemental or alternative therapy during the baseline or treatment phases of the clinical study. This includes: acupuncture, spinal manipulation, TENS, and magnetic field treatments.
12. Subject agrees to maintain current preventative headache medication regimens (no change in type, frequency, or dose) from baseline screening visit to the end of the Phase 2 treatment phase.

Exclusion Criteria:

1. Subject currently has Medication Overuse Headache (MOH) in the judgment of the investigator or by ICHD-II criteria.
2. Subject has a history of headaches days ≥ 15 per month.
3. Subject has a history of trigeminal autonomic cephalalgias.
4. Subject has any medical condition or disorder that:

   1. Is considered to be clinically significant and may pose a safety concern
   2. Could interfere with the accurate assessment of safety or efficacy
   3. Could potentially affect a subject's safety or study outcome.
5. Subject has had a major infection or surgery in the past month.
6. Subject has undergone facial surgery in the area of sphenopalatine ganglia for cosmetic, corrective, therapeutic, or traumatic reasons.
7. Subject has been treated with radiation to the face.
8. Subject was diagnosed with any major infectious processes, primary or secondary malignancies involving the face that have been active or required treatment in the past six (6) months.
9. Subject currently meets criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) for an active major depressive episode or for active significant psychiatric disorders, including dementia, uncontrolled general anxiety disorder, psychotic disorders or uncontrolled bipolar disorder. Exclusion criteria include: suicidality, active psychosis, untreated severe depression and/ or anxiety disorder, litigation, addiction, homicidal ideation, significant Axis II disorders and untreated sleep disorder.
10. Subject currently has clinically significant drug or alcohol abuse as defined by DSM-IV-TR or is unable to refrain from substance abuse throughout the study.
11. Subject is currently participating or has participated in the last month in another clinical study in which the subject has, is, or will be exposed to an investigational or non-investigational drug or device.
12. Subject is felt to be at risk of non-compliance (e.g. for completing the diary or maintaining a stable headache medicine regimen) in the investigator's opinion.
13. Subject is woman of childbearing age who is pregnant, nursing, or not using contraception.
14. Subject has had previous radio-frequency ablation of the SPG.
15. Subject has had blocks of the SPG in last 3 months.
16. Subject has undergone botulinum toxin injections of the head and/or neck in the last 3 months.
17. Subject has an implantable stimulator or any implanted devices in the head and/or neck.
18. Subject has H/O bleeding disorders or coagulopathy, or is on anticoagulation, antiplatelet, or GP IIb IIIa inhibitor medication.
19. Subject has H/O malignancy or any other condition that requires MRI monitoring.
20. Subject has or requires pacemaker/defibrillator.
21. Subject is not suitable for the study, in the judgment of the Investigators, due to social, co-morbid psychological, and/or medical considerations.
22. Subject has H/O stroke, cardiovascular disease, and/or epilepsy.
23. Subject was on antipsychotic or antidepressant medications (except for migraine prevention) in the past 3 months prior to the study.
24. Subject is allergic or has shown hypersensitivity to materials of the Medtronic components which come in contact with the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Tepper, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol required 3 subjects who were from the Cleveland Clinic migraine patient population.
Pre-assignment Details: This is a one arm study
Groups:
- Deep Brain Stimulation Arm Group: Electrical Stimulation of SPG for Treatment of Migraine
  Electrical Stimulation of SPG for Treatment of Migraine: Electrical Stimulation of the Sphenopalatine Ganglion for the Treatment of Migraine Headaches
Period: Overall Study
Arm/Group | Deep Brain Stimulation Arm Group
Started | 3
Completed | 0
Not Completed | 3
Not completed — Infection and surgical explant | 1
Not completed — Eligibility criteria expanded | 1
Not completed — Stimulation response inadqequate | 1

BASELINE CHARACTERISTICS:
Population: no subjects had data collected, 3 were enrolled, but did not have data collected or analyzed.
Arm/Group | Deep Brain Stimulation Arm Group
Number analyzed (Participants) | 0
Age, Categorical
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Migraine Relief at 2 Hours Post Stimulation
Description: Pain is rated at stimulation and 2 hours after stimulation initiated based on four point categorical scale, FDA-approved, where 0 = no headache pain, 1= mild pain, 2 = moderate pain, 3 = severe pain. This scale has been used since 1991 for all regulatory submission migraine protocols. Each migraine is categorized in a binary fashion as meeting the endpoint at 2 hours. Migraine relief or Pain relief is defined as moving from pain levels of 3 to 2 down to 1 or 0.
Time Frame: 8.5 Months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation Arm Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Migraine Free at 2 Hours
Description: Each migraine will be categorized as meeting the endpoint of migraine free if there is a reduction in the migraine grade to 0 for pain with no nausea, photophobia and phonophobia at 2 hours after initiation of stimulation.
Time Frame: 8.5 Months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation Arm Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Free at 2 Hours Post Stimulation
Description: As noted above, we are using the FDA-approved categorical scale used for all migraine regulatory trials since 1992. This is a 4 point categorical scale where 0= no pain, 1= mild headache pain, 2= moderate pain, and 3= severe pain. Pain free is defined as the subject moving from pain intensity of 2 to 3 at baseine to 0 by 2 hours after stimulation.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Groups:
- Experimental: Deep Brain Stimulation Arm Group: Experimental: Deep brain stimulation arm group
  Electrical Stimulation of SPG for Treatment of Migraine
Arm/Group | Experimental: Deep Brain Stimulation Arm Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Acute Migraine Medication Use
Description: During the baseline period, subjects will record their acute as-needed migraine relief medication use for each attack by drug, dose, route, and frequency. A secondary endpoint for this phase is a reduction in acute migraine medication usage for each attack for drug, dose, route, and frequency during the last month of the study as compared to the baseline month.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Groups:
- Deep Brain Stimulation of SPG for Migraine: Electrical SPG for Treatment of Migraine
  Deep Brain Stimulation of SPG for Migraine: Deep Brain Stimulation of SPG for Migraine
  No outcome measure data was analyzed because no outcome data were collected.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

5. Secondary Outcome: Headache Impact Test (HIT-6) Compared With Baseline
Description: The Headache Impact Test -6 (HIT-6) is a validated tool for evaluating headache impact and disability across 6 domains, which will be recorded at baseline and at study conclusion.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation Arm Group
Number analyzed (Participants) | 0

6. Secondary Outcome: Migraine Disability Assessment Scale (MIDAS) at Study Conclusion Compared With Baseline
Description: The Migraine Disability Assessment Scale (MIDAS) is a validated tool that assesses how many days in the last 3 months a patient had at least 50% disability at work, home, school, or recreational activities due to migraine. MIDAS will be assessed at baseline and after study conclusion.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Groups:
- Deep Brain Stimulation of SPG for Migraine: Electrical SPG for Treatment of Migraine
  Deep Brain Stimulation of SPG for Migraine: Deep Brain Stimulation of SPG for Migraine
  No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

7. Secondary Outcome: Stimulation Related Adverse Events
Description: Number of Participants with Adverse Events as a Measure of Safety and Tolerability
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

8. Secondary Outcome: Average Per Subject Reduction in Migraine Days/Month
Description: During the baseline period, subjects will record the number of migraine days (as defined by the FDA-approved International Classification of Headache Disorders, 2d Edition definition of migraine with and without aura) during the month. The primary endpoint for this phase is a reduction in the number of migraine days during the last month of the study as compared to the baseline month.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

9. Secondary Outcome: Implantation and Stimulation Related Adverse Events
Description: as for outcome 3
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

10. Secondary Outcome: Relief of Migraine-associated Symptoms, e.g. Nausea/Vomiting, Photophobia, Phonophobia
Description: Presence or absence of nausea, vomiting, photophobia, and phonophobia will be assessed at baseline and after stimulation at 2 hours for each stimulation for each individual.
Time Frame: 8.5 months
Population: No data were collected from this entire study, so no data were analyzed.
Arm/Group | Deep Brain Stimulation of SPG for Migraine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month, the time between implant and explant which was performed due to subject infection. No treatment period occurred.
Description: There was one adverse event which was an infection which required the explant surgery. Full report was made to the FDA and the IRB of this adverse event.
  The other two subjects who were consented and enrolled did not receive any treatment and no adverse events were noted.
Arm/Group | Deep Brain Stimulation Arm Group
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation Arm Group (N=1)
Infection and surgical explant (Nervous system disorders) | 1 (1) — Infection and surgical explant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes